CLINICAL TRIAL: NCT05895747
Title: 31P-MRS and Resting State Functional Connectivity Analysis of the Effects of 5-hydroxytryptophan and Creatine for Antidepressant Augmentation in Patients With SSRI/SNRI-resistant Major Depressive Disorder
Brief Title: 5-HTP and Creatine for Depression R33 Phase
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Brent Michael Kious, MD, PhD, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB_00132830_R33
Record Dates: First submitted 2023-05-25; First posted 2023-06-09 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — 5-Hydroxytryptophan; Creatine; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low Dose 5-hydroxytryptophan and Creatine Monohydrate (Experimental): 5-HTP 100mg PO BID plus creatine 5g PO Qday
  Interventions: Drug: Low Dose 5-hydroxytryptophan; Drug: Low Dose Creatine Monohydrate; Drug: Placebo
- High Dose 5-hydroxytryptophan and Creatine Monohydrate (Experimental): 5-HTP 200mg PO BID plus creatine 10mg PO Qday
  Interventions: Drug: High Dose 5-hydroxytryptophan; Drug: High Dose Creatine Monohydrate
- Double Placebo (Placebo Comparator): Creatine-matched placebo and 5-HTP-matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low Dose 5-hydroxytryptophan — 5-hydroxytryptophan 100mg PO BID
  Other Names: 5-HTP
  Arms: Low Dose 5-hydroxytryptophan and Creatine Monohydrate
Drug: High Dose 5-hydroxytryptophan — 5-hydroxytryptophan 200mg PO BID
  Other Names: 5-HTP
  Arms: High Dose 5-hydroxytryptophan and Creatine Monohydrate
Drug: Low Dose Creatine Monohydrate — Creatine monohydrate 5g PO qday
  Other Names: creatine
  Arms: Low Dose 5-hydroxytryptophan and Creatine Monohydrate
Drug: High Dose Creatine Monohydrate — Creatine monohydrate 10g PO qday
  Other Names: creatine
  Arms: High Dose 5-hydroxytryptophan and Creatine Monohydrate
Drug: Placebo — Creatine-matched placebo and 5-HTP-matched placebo; Placebo will be dextrose either encapsulated (5-HTP matched) or as loose powder (creatine matched)
  Other Names: dextrose
  Arms: Double Placebo; Low Dose 5-hydroxytryptophan and Creatine Monohydrate

SUMMARY:
This is a three-armed clinical trial examining the effect of 5-hydroxytryptophan and creatine monohydrate as augmenting agents for the treatment of depression. Subjects will be randomized between 5-HTP 100mg BID + creatine 5g daily, 5-HTP 200mg BID + creatine 10g daily, vs double placebo, for 8 weeks. The ability of the interventions to affect biomarkers associated with depression will be assessed using brain phosphorus magnetic resonance spectroscopy, functional connectivity imaging, and plasma serotonin levels.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) has a lifetime prevalence of over 16% and is associated with reduced work productivity, disability, increased mortality, and increased rates of suicide attempts and completed suicides. Unfortunately, ~34% fail to respond to standard ADs (ADs). Environmental and patient-level factors that increase the risk of MDD could pinpoint novel mechanisms underlying the disorder. One such factor may be relative hypoxia. Persons with hypoxic medical conditions, such as asthma and chronic obstructive pulmonary disease, are at higher risk of depression and suicide compared to those with other chronic medical conditions. Smoking also promotes hypoxia and is linked to increased risks of suicide and depression. Of special relevance to this study, living at high altitude produces relative hypoxia even after months, and is linked to increased risks of suicide and depression. Hypoxia could contribute to MDD in at least two ways. First, brain bioenergetics are altered in both hypoxia and MDD. Hypoxia reduces several neurochemical markers of brain activity, including phosphocreatine (PCr) and n-acetylaspartate (NAA), and alters mitochondrial dynamics in the hippocampus. Proton magnetic resonance spectroscopy (1H-MRS) shows that high-altitude residents have altered whole brain pH and reduced inorganic phosphate to total phosphate (tP) ratios compared to persons dwelling at sea-level. In depressed patients, phosphorus MRS (31P-MRS) shows reduced nucleotide triphosphate (NTP) concentrations and decreased PCr concentrations; AD response is associated with increases in PCr and NTP. Hypoxia could also promote MDD by altering serotonin (5-HT) production. Chronic hypoxia reduces 5-HT in the forebrain and brainstem in rodents. The conversion of tryptophan to 5-hydroxytryptophan (5-HTP) by tryptophan hydroxylase is oxygen-dependent and slowed by hypoxia. Animal studies have shown that selective serotonin reuptake inhibitors (SSRIs) are not as effective at altitude, possibly because of inadequate 5-HT production. Reductions in 5-HT synthesis and inefficiencies in bioenergetics could both contribute to altered brain functional connectivity. MDD may disrupt cortical emotion regulation, and resting state functional connectivity (fcMRI) studies suggest that depression involves reduced connectivity between frontal cortical regions and the amygdala, while AD response correlates with normalization of those connections. Alterations in connectivity associated with AD response are correlated with changes in brain metabolites, suggesting a link to brain bioenergetics.

This suggests two natural supplements as interventions for depression. Oral creatine monohydrate (Cr) could improve bioenergetics in MDD, as Cr alters brain tCr, PCr, and NTP levels. Moreover, Cr produces improvements in mood correlated with normalization of PCr levels and structural connectivity. Alterations in 5-HT synthesis due to hypoxia could be rectified by 5-HTP, as its conversion to 5-HT is not oxygen-dependent. 5-HTP elevates brain 5-HT levels and has AD efficacy in clinical trials. The proposed study is a two-phase, three-armed trial to evaluate whether SSRI/SNRI augmentation with the supplements Cr, 5-HTP, or their combination (5-HTP+Cr) can enhance AD response in treatment-resistant MDD. In the R61 phase, the study will assess the ability of the interventions to alter biological signatures associated with depression, as measured by 31P-MRS, fcMRI, and changes in whole blood 5-HT. In the R33 phase, the study will attempt to replicate the above findings with dose variation and evaluate their correlation with clinical outcomes. The study will have the following aims:

Aim 1. Replicate the clinically meaningful changes in biological signatures (PCr:tP ratios as measured by 31P-MRS, sgACC connectivity as measured by fcMRI, and whole blood serotonin) demonstrated in the R61 phase, following the decision rule noted above.

Aim 2. Demonstrate that the changes in each of the above markers that is carried over from the R61 phase are correlated with changes in depression as measured by the 17-item Hamilton Depression Rating Scale, which would be studied in a subsequent efficacy trial.

Study results will help elucidate the potential efficacy of a novel combination of nutritional supplements in persons with MDD, given strong epidemiologic and physiologic evidence suggesting that relative hypoxia can contribute to depression through alterations in brain bioenergetics and 5-HT synthesis. Target engagement will be indicated by improvements in functional connectivity and frontal cortical energy metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18-65 years inclusive
* Current diagnosis of MDD identified by the MINI (Mini Neuropsychiatric Interview)
* Current HAM-D17 score of >= 16
* Adequate adherence to any FDA approved SSRI or SNRI for at least 8 weeks
* Right-handed
* Residing at > 4000 ft for at least 12 weeks

Exclusion Criteria:

* Any non-MDD and non-anxiety psychiatric diagnosis, as identified by the MINI
* History of or current diagnosis of renal disease, such as chronic renal failure, acute renal failure or end stage renal disease
* Current colitis or diverticulitis
* History of or current pulmonary disease (except well controlled asthma)
* Current smoking
* History of cardiac disease or QTc > 500ms
* History of fibromyalgia or any rheumatological condition
* History of or current seizure disorder
* Current serious suicide risk identified by the Columbia Severity Suicide Rating Scale
* Current treatment with an antipsychotic, mood stabilizer, or non-SSRI/SNRI antidepressant except for bupropion at FDA-approved doses or trazodone up to 200mg, or use of any supplements apart from standard multivitamins
* Positive pregnancy test, pregnancy, failure to use adequate birth control method
* Previous diagnosis of serotonin syndrome or evidence of serotonin syndrome
* Pre-existing eosinophilia (absolute eosinophil count > 500/uL)
* Contraindications to MRI: ferromagnetic implants, implanted devices, claustrophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
17-Item Hamilton Depression Rating Scale | 8 weeks
  Hamilton Depression Rating Scale response: >=50% reduction in baseline score; maximum possible score is 52, minimum possible score is 0. Higher scores suggest more severe depression.

SECONDARY OUTCOMES:
Montgomery Asberg Depression Rating Scale | 8 weeks
  Montgomery Asberg Depression Rating Scale; Response is a >=50% reduction in baseline score; minimum score 0; maximum score 60; higher scores suggest more severe depression

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah Department of Psychiatry, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No